CLINICAL TRIAL: NCT01340859
Title: Inpatient Post Admission Cognitive Therapy (PACT) for the Prevention of Suicide Attempts: A Pilot Study
Brief Title: Inpatient Post Admission Cognitive Therapy (PACT) for the Prevention of Suicide Attempts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Principal Investigator, Marjan Holloway, Associate Professor, Henry M. Jackson Foundation for the Advancement of Military Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: G172JF
Record Dates: First submitted 2011-04-21; First posted 2011-04-25 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Suicide, Attempted
Keywords: Suicide; Cognitive Therapy; Inpatient; Military
MeSH Terms: conditions — Suicide, Attempted; Suicide | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Post Admission Cognitive Therapy (PACT) (Experimental): Six (6) 60-90 Minutes Sessions of Post Admission Cognitive Therapy Delivered Preferably Over 3 Consecutive Days of Inpatient Stay
  Interventions: Behavioral: Post Admission Cognitive Therapy (PACT)
- Enhanced Usual Care (EUC) (No Intervention): Treatment As Usual and Study Assessment Services

INTERVENTIONS:
Behavioral: Post Admission Cognitive Therapy (PACT) — Individual psychotherapy; 60-90 minutes sessions; 6 sessions over preferably 3 days of inpatient stay
  Other Names: Cognitive Therapy; Cognitive Behavior Therapy
  Arms: Post Admission Cognitive Therapy (PACT)

SUMMARY:
The broad objective of this research is to effectively utilize a unique window of opportunity during the hospitalization period following a recent suicide attempt to deliver a brief and targeted intervention for suicidal individuals.

DETAILED DESCRIPTION:
Suicide remains a serious public health problem as the 4th leading cause of death among individuals 15-44 years old and the 2nd leading cause of death in the military. Developing effective interventions for suicide behavior has been a stated goal of the National Strategy for Suicide Prevention. To date, only a limited number of controlled studies have examined the efficacy of psychosocial interventions in reducing suicide behavior. Preliminary findings from the University of Pennsylvania (Brown et al., 2005) indicate that outpatient cognitive therapy reduces the likelihood of repeat suicide attempts by approximately 50%. Yet the efficacy of this promising new intervention has not been tested in other medical settings or in other specific at risk groups.

We propose an adaptation of Beck and colleagues cognitive therapy suicide protocol for implementation, feasibility, and pilot testing at an inpatient psychiatry setting for specific delivery to military service members and their family members with a recent suicide attempt. Suicide attempt behavior is one of the most powerful risk factors for repeat suicide behavior as well as eventual death by suicide. Delivering a brief and possibly potent psychotherapeutic intervention during a patient's inpatient hospitalization aims to directly target individuals at high risk for future suicide behavior, i.e., young adult, mostly males with a recent suicide attempt, under direct stress of a military career. We expect that the adapted intervention, titled Post Admission Cognitive Therapy (PACT), will show promise in reducing the likelihood of post-hospitalization suicide attempt behavior as well as psychological risk factors associated with suicide such as depression, hopelessness, suicide ideation, and posttraumatic symptoms. Our proposed design is a randomized controlled pilot trial with blinded outcome assessments.

Specific Aims: (1) To develop and evaluate a new manual of Post-Admission Cognitive Therapy (PACT) as a targeted inpatient treatment for individuals admitted for a recent suicide attempt to a military hospital. (2) To assess the feasibility of the study's assessment procedures by monitoring the completion rate of outcome measures during face-to-face as well as follow-up phone and web-based administrations. (3) To evaluate the degree of change and variability of response to Post-Admission Cognitive Therapy in comparison to Enhanced Usual Care at post-intervention and follow-up (1-, 2-, and 3-Month) on subsequent suicide attempt behavior (primary outcome) as well as on levels of depression, hopelessness, and suicide ideation (secondary outcomes). (4) To examine in a preliminary manner whether improvements on primary and secondary outcome measures are associated with enhanced problem solving abilities which is viewed as a potential mechanism of change in cognitive therapy for the reduction of suicide behavior.

Study Design: We plan to randomize 24 patients hospitalized at the Walter Reed National Military Medical Center for a recent suicide attempt to one of two conditions: (1) Post-Admission Cognitive Therapy + Enhanced Usual Care (PACT+EUC) or (2) Enhanced Usual Care (EUC). Individuals who are over the age of 18, able to communicate in English and willing to provide informed consent will be recruited. The PACT+EUC condition will consist of six 60-90 minute individual cognitive therapy sessions administered preferably over 3 days. The EUC condition will consist of the usual care patients receive at an inpatient facility during their hospitalization in addition to assessment services provided by independent evaluators who work directly with our research team. The primary outcome variable is the number of subsequent suicide attempts. We expect that patients in the control condition will reattempt suicide at an earlier date and at a higher frequency as compared to patients enrolled in the intervention condition. Secondary outcome measures include the severity of depression, hopelessness, and suicide ideation. Patients in both conditions will be assessed on the dependent measures at baseline and at 1-, 2-, and 3- month follow-up intervals. Data analyses will provide estimates of the statistical power of PACT relative to EUC over time via the usage of repeated observation data. Our preliminary effect size estimates will be used for future sample size calculations to conduct a larger randomized controlled trial to definitively determine the efficacy of PACT.

ELIGIBILITY:
Inclusion Criteria:

* Recent Suicide Attempt
* Baseline Completed Preferably within 48 Hours of Admission
* Over the Age of 18
* Provides Informed Consent

Exclusion Criteria:

* Self-Inflicted Harm with No Intent or Desire to Die
* Medical Incapacity to Participate
* Current State of Active Psychosis
* Expected Discharge within 72 Hours of Admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-04; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Repeat Suicide Attempts | 1, 2, and 3 months
  Columbia Suicide Severity Rating Scale; Hospital Records

SECONDARY OUTCOMES:
Depression | 1, 2, and 3 months
  Beck Depression Inventory
Hopelessness | 1, 2, and 3 months
  Beck Hopelessness Scale
Suicide Ideation | 1, 2, and 3 months
  Scale for Suicide Ideation and Columbia Suicide Severity Rating Scale
Post-Traumatic Stress Symptoms | 1, 2, and 3 months
  Various measures on trauma
Reliable Change Index | 1, 2, and 3 months
  Clinical change that can be considered as meaningful

CONTACTS AND LOCATIONS:
Overall Officials: Marjan G Holloway, Ph.D., Principal Investigator — Uniformed Services University of the Health Sciences
Locations (2):
- United States (2):
  - Uniformed Services University of the Health Sciences, Bethesda, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghahramanlou-Holloway M, Cox D, & Greene F. Post-admission cognitive therapy: A brief intervention for psychiatric inpatients admitted after a suicide attempt. Cognitive and Behavioral Practice 19: 233-244, 2012.
- [Background] Kochanski-Ruscio KM, Carreno-Ponce JT, DeYoung K, Grammer G, Ghahramanlou-Holloway M. Diagnostic and psychosocial differences in psychiatrically hospitalized military service members with single versus multiple suicide attempts. Compr Psychiatry. 2014 Apr;55(3):450-6. doi: 10.1016/j.comppsych.2013.10.012. Epub 2013 Nov 4. PMID 24387921
- [Derived] LaCroix JM, Colborn VA, Hassen HO, Perera KU, Weaver J, Soumoff A, Novak LA, Ghahramanlou-Holloway M. Intimate partner relationship stress and suicidality in a psychiatrically hospitalized military sample. Compr Psychiatry. 2018 Jul;84:106-111. doi: 10.1016/j.comppsych.2018.04.006. Epub 2018 Apr 21. PMID 29747068